CLINICAL TRIAL: NCT00198367
Title: Three Modalities of Treatment in Operable and Resectable Stage IIIA (T1-3, N2) NSCLC. Randomized Phase II Study
Brief Title: Three Modalities of Treatment in Operable and Resectable Stage IIIA (T1-3, N2) Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-0101
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2016-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: operable and resectable stage IIIA (T1-3, N2) NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

ARMS (3):
- Cisplatin-Gemzar (Experimental): Cisplatin-Gemzar
  Interventions: Drug: Cisplatin-Gemzar
- Cisplatin-Navelbine-Radiotherapy (Experimental): Cisplatin-Navelbine-Radiotherapy
  Interventions: Drug: Cisplatin-Navelbine-Radiotherapy
- Carboplatin-Taxol-Radiotherapy (Experimental): Carboplatin-Taxol-Radiotherapy
  Interventions: Drug: Carboplatin-Taxol-Radiotherapy

INTERVENTIONS:
Drug: Cisplatin-Gemzar
  Arms: Cisplatin-Gemzar
Drug: Cisplatin-Navelbine-Radiotherapy
  Arms: Cisplatin-Navelbine-Radiotherapy
Drug: Carboplatin-Taxol-Radiotherapy
  Arms: Carboplatin-Taxol-Radiotherapy

SUMMARY:
Stage IIIA non-small cell lung cancers comprising a mediastinal ganglionic invasion N2 account for 20 to 30% of the NSCLCs. They are almost always potentially resectable, but the results obtained by surgery alone or surgery followed by chemotherapy (CT) and/or radiotherapy (RT) are insufficient. The neoadjuvant approach was tested, in randomized tests of exclusive CT, or in noncomparative tests of RT-CT.

DETAILED DESCRIPTION:
These results justify the choice of the study design currently suggested, testing the preoperative feasibility

1. chemotherapy: cisplatin-Gemzar (arm A) or
2. chemoradiotherapy: cisplatin-navelbine-radiotherapy (arm B) or Carboplatin-Taxol-radiotherapy (arm C).

The results obtained, in terms of feasibility and toxicity, will make it possible to select the optimal diagrams for a phase III study.

ELIGIBILITY:
Inclusion Criteria:

* Operable and resectable stage IIIA (T1-3, N2) NSCLC
* World Health Organization (WHO) performance status of 1 or less

Exclusion Criteria:

* Severe cardiac, respiratory, renal or hepatic failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2003-01; Primary Completion 2008-01 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
percentage of patients alive and operated on without grade 4 toxicity (except for hematological and N/V toxicities) | at week 22

CONTACTS AND LOCATIONS:
Overall Officials: Francoise Mornex, Pr, Principal Investigator — Hospices Civils de Lyon; Bernard Milleron, Dr, Principal Investigator — Intergroupe Francophone de Cancerologie Thoracique
Locations (1):
- Centre Hospitalier Lyon-Sud - Radiotherapie/Oncologie, Pierre-Bénite, France

REFERENCES:
- [Result] Girard N, Mornex F, Douillard JY, Bossard N, Quoix E, Beckendorf V, Grunenwald D, Amour E, Milleron B. Is neoadjuvant chemoradiotherapy a feasible strategy for stage IIIA-N2 non-small cell lung cancer? Mature results of the randomized IFCT-0101 phase II trial. Lung Cancer. 2010 Jul;69(1):86-93. doi: 10.1016/j.lungcan.2009.10.003. Epub 2009 Oct 29. PMID 19879013